CLINICAL TRIAL: NCT05084027
Title: Venetoclax Combining With Fludarabine and Melphalan as Conditioning Regimen Prior to Allogeneic Hematopoietic Stem Cell Transplantation for Older Patients With Hematologic Malignancies
Brief Title: Venetoclax Combining With Fludarabine and Melphalan as Conditioning Regimen for Allo-HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Zhejiang Provincial People's Hospital (Other); The Affiliated People's Hospital of Ningbo University (Other Government); First Affiliated Hospital of Wenzhou Medical University (Other); Ningbo Hospital of Zhejiang University (Unknown); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Yi Luo, Principal Investigator, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJU-HSCT-RIC
Record Dates: First submitted 2021-10-07; First posted 2021-10-19 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Hematologic Malignancy; Older Patients; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fludarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): older patients accepting venetoclax combining with fludarabine and melphalan as conditioning regimen prior to allogeneic hematopoietic stem cell transplantation treatment
  Interventions: Combination Product: venetoclax combining with fludarabine and melphalan

INTERVENTIONS:
Combination Product: venetoclax combining with fludarabine and melphalan — Venetoclax 400mg/day，oral，day-8～day-2; Fludarabine, 30mg/m2/day，intravenous，d-7～d-3；Melphalan, 140mg/ m2/d，intravenous，day-2

SUMMARY:
venetoclax combining with fludarabine and melphalan as conditioning regimen prior to allogeneic hematopoietic stem cell transplantation for older patients with hematologic malignancies

DETAILED DESCRIPTION:
It was a phase Ⅱ clinical trial of new designed reduced-intensity conditioning regimen for older patients accepting allogeneic hematopoietic stem cell transplantation treatment. The regimen consisted of venetoclax combining with fludarabine and melphalan.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 50 years
2. Patients diagnosed with acute myeloid leukemia, acute lymphoblastic leukemia, myelodysplastic syndrome according to WHO diagnostic criteria.
3. Patients who achieved complete remission before transplantation.
4. Patients who have alternative donors and plane to accept allogeneic hematopoietic stem cell transplantation treatment.
5. ECOG body status score 0-2.
6. Good organ function level: ANC (neutrophil absolute value >=1.0x10^9/L; PLT >=30x10^9/L; HB >=80g/L; Tibil <=1.5 ULN; ALT / AST <=2.5 ULN; bun / Cr <=1.5 ULN; LVEF >=50%).
7. Patients who voluntarily participate in the clinical trial, understand the research procedure and can sign the informed consent in writing.

Exclusion Criteria:

1. Patients who didn't achieved complete remission before transplantation (bone marrow smear: proportion of primordial cells >=5%) or any extramedullary recurrence.
2. Patients who were previously known to be resistant to venetoclax.
3. In patients with severe pulmonary insufficiency (obstructive and / or restrictive ventilation disorders), the researchers evaluated the patients who could not tolerate the super pretreatment scheme.
4. Patients with severe liver function impairment and liver function indexes (alt, TBIL) more than 3 ULN were evaluated as intolerant of super pretreatment.
5. In patients with severe renal insufficiency, the renal function index (CR) is more than 2 times of the upper limit of the normal value (ULN), or the 24-hour creatinine clearance rate (CR) is less than 50ml / min, the researchers evaluated that they could not tolerate the super pretreatment scheme.
6. In patients with severe active infection, the researchers evaluated that they could not tolerate the pretreatment.
7. Patients who had allergic reactions or serious adverse reactions in the previous use of pretreatment related drugs could not be included in the study.
8. Other reasons why the researchers could not be selected.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 2 year
  2-year DFS

SECONDARY OUTCOMES:
incidence of toxic reaction | 2 year
  2-year incidence of toxic reaction
overall survival | 2 year
  2-year OS
cumulative incidence of relapse | 2 year
  2-year incidence of relapse
incidence of acute and or chronic graft verus host disease | 2 year
  2-year incidence of cGVHD

CONTACTS AND LOCATIONS:
Overall Officials: Yi Luo, M.D., Principal Investigator — First Affilaated Hospital of Medical School of Zhejiang University
Locations (8):
- China (8):
  - The first Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - First Affiliated Hospital of Zhejiang Chinese Medicine University, Hangzhou, Zhejiang
  - Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, College of Medicine, Zhejiang University, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Ningbo Hospital of Zhejiang University, Ningbo
  - The Affiliated People's Hospital of Ningbo University, Ningbo
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou

IPD SHARING:
Plan to Share IPD: No